CLINICAL TRIAL: NCT04502329
Title: The Effect of Intermittent Fasting Diet on Metabolic Syndrome Biomarkers and Weight Management in Individuals With Metabolic Syndrome
Brief Title: Does the Energy Restriction Intermittent Fasting Diet Alleviate Metabolic Syndrome Biomarkers?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, yaseminkunduraci, Clinical Dietitian, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10840098-604.01.01-E.1866
Record Dates: First submitted 2020-06-15; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Metabolic Syndrome
Keywords: intermittent fasting; metabolic syndrome; time restricted diet; energy restriction
MeSH Terms: conditions — Metabolic Syndrome; Intermittent Fasting | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Randomized control trial The first participant assigned Intermittent Energy Restriction Group, the others assigned Continous Energy Restricition group or Intertermittent Energy Restriction Group respectively.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IER (Experimental): Intermittent Energy Restriction
  Interventions: Other: Diet
- CER (No Intervention): Continous Energy Restriction

INTERVENTIONS:
Other: Diet — Energy Restriction Intermittent Fasting Diet
  Arms: IER

SUMMARY:
The aim of this randomized controlled study determine the efficacy of calorie restriction intermittent fasting diet in metabolic parameters and weight management among metabolic syndromes adults. It was done on metabolic syndrome patients, aged 18-65 years at an academic institution in Istanbul,Turkey. Subjects were divided into two groups; IER (Intermittent Energy Restriction-intervention group, calori restriction of 300-500kcal/d combined with 16:8 model Intermittent Fasting) and CER (Countinous Energy Restriction- control group continous restriction of 300-500kcal/d). Assessment was ascertained at baseline and 12 weeks. Blood samples were analyzed for lipid profile, fasting plasma glucose, ınsulin, HOMA-IR. Blood pressure and body composition were evaluated.

DETAILED DESCRIPTION:
Aim The aim of this study; determine the efficacy of calorie restriction intermittent fasting diet in metabolic parameters and weight management among metabolic syndromes adults.

Subjects Participants who referred by clinician, as medical doctors after physical assesment selected in this study were recruited among patients with metabolic syndrome referring to the diet clinic local in Turkey. The criteria of inclusion were metabolic syndrome patients, aged 18-65 years had body mass index (BMI) ≥27 kg/m2 with no history of mental or physical disabilities.Subjects should also not be practicing Muslim Ramadan fasting or had changed their dietary pattern 12 weeks before the study. Eligible subjects were approached to participate. Only those who agreed to participate were explained of all the information pertaining to this study and were consented. This study was approved by Istanbul Medipol University Ethics Committee.

Study design The aim of A randomized controlled study was carried out to determine the efficacy of calorie restriction intermittent fasting diet in metabolic parameters and weight management among metabolic syndromes adults. Subjects were randomly assigned into two groups; intervention IER (Intermittent Energy Restriction) and control CER (Continuous Energy Restriction). Randomization, first participant assigned IER group an each eligible participant was randomly assigned to either CER group or IER group. Those who were assigned to two groups needed to adhere dietary regime, with a reduction of 300-500kcal/d from the habitual energy intake for 12 weeks intervention period. Diet menus were prepared taking into account the individual characteristics. IER participants abide by intermittent fasting which time restricted 16:8 model diet. During 16 hours; such as at 04.00 pm- 08.00 am or 05.00 pm - 09.00 am or 07.00 pm - 11.00 am fasting hours, no food and calorie drink. But participants in fasting hours can drink water, sugar free tea and mineral water, coffee without sauce. On the other 8 hours, need to adhere energy restriction diet. Subjects were also provided with seven-day food menu guidelines. Those who were assigned to two groups need to maintain their present lifestyle. Analysis was carried out at two time points: baseline and week 12. In order to ensure good compliance, subjects were contacted once a week via telephone calls. Food diaries and were fasting log book presumed to the participants during each assessment meeting. Subjects were given detailed instruction verbally and a reference guide on how to fill up the food diaries and fasting log. Individual and group counseling were provided before and during the intervention period.

Body composition, Blood Pressure, Biochemical markers Height was measured using SECA-213 portable stadiometer (SECA, Hamburg, Germany). Body composition was measured using TANITA SC-330, body composition analyzer (TANITA Corp. Tokyo, Japan). All measurements were made in the morning at participants fasted state. This instrument was calibrated each time before measurement. Data from this instrument including body weight, BMI, body fat percentage, fat mass, fat free mass and total body water.

Body mass index (BMI) was calculated as; BMI [kg/m2]= Weight[kg] / (Height[m] x Height[m]) Waist circumference was measured by the same dietician with the help of a standard unstretched tape measure. Blood pressure and heart rate were measured using an automatic oscillometric device (Omron M2 Basic, Japanese) after participants had rested in a seated position for 5 min. A blood sample was drawn at baseline and after 12 weeks. Insulin resistance was estimated with the homeostasis model assessment (HOMA-IR) and calculated as; HOMA-IR= (Fasting plasma glucose [mg/dL] x Serum insulin [IU/L]) / 405

Biochemical markers blood lipids, fasting plasma glucose and Haemoglobin A1c (HbA1c) were performed with standard methods. Serum concentrations of insulin were measured by immunonephelometric methods. Adverse events were monitored by standardized questionnaires, diary and at the last study visit by interview.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Body mass index to be 27 and above
* Clinical diagnosis of metabolic syndrome according to the criteria of IDF 2005 or NCP ATP III.

Exclusion Criteria:

* Being in the pre-menopausal or menopause
* Following a special diet (such as Celiac, Type 1 diabetes)
* Using a special nutritional supplement (omega 3, probiotic, vitamin-mineral, teff seed etc.)
* Those who do not comply with the diet, pregnant, being lactating
* Doing heavy physical activity or working in a heavy job
* Presence of liver, kidney or immune deficiency
* Conditions that will seriously affect weight management such as having bariatric surgery
* Determined to have had an unintentional sudden weight loss of more than 5% in the last three months
* Not be practicing Muslim Ramadan fasting or had changed their dietary pattern 12 weeks before the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Average weight and standard deviation of the participants | Change from Baseline Weight at 12 weeks
  Weight in kilograms, was measured with TANİTA SC-330 instrument.
Average height and standard deviation of the participants | Baseline
  Height measured with SECA-213 instrument.
Average Body Mass Indexand standard deviation of the participants | Change from Baseline Body Mass Index at 12 weeks
  Weight and Height were combined to report BMI in kg/m^2
Average Waist circumference and standard deviation of the participants | Change from Baseline Weight at 12 weeks
  Waist circumference in centimeters, was measured by the same dietician with the help of unstretched tape measure.
Concentration of Total Cholesterol | Change from Baseline Weight at 12 weeks
  Total cholesterol in mg/dL, results was provided from participant's clinician before and 12 weeks after diet.
Concentration of High-Density Cholesterol | Change from Baseline Weight at 12 weeks
  High Dansity Cholesterol in mg/dL, results was provided from participant's clinician before and 12 weeks after diet.
Concentration of Low-Density Cholesterol | Change from Baseline Weight at 12 weeks
  Low Dansity Cholesterol in mg/dL, results was provided from participant's clinician before and 12 weeks after diet.
Concentration of Triglyceride | Change from Baseline Weight at 12 weeks
  Triglyceride in mg/dL, results was provided from participant's clinician before and 12 weeks after diet.
Concentration of Fasting plasma glucose | Change from Baseline Weight at 12 weeks
  Fasting plasma glucose in mg/dL, was provided from participant's clinician before and 12 weeks after diet.
Concentration of Insülin | Change from Baseline Weight at 12 weeks
  Insülin in IU/L, was provided from participant's clinician before and 12 weeks after diet.
Rate of HOMA-IR | Change from Baseline Weight at 12 weeks
  HOMA-IR was calculated with fasting plasma glucose and insülin levels. HOMA-IR = (Fasting plasma glucose [mg/dL] x Insülin [IU/L] ) / 405
Concentration of HbA1c | Change from Baseline Weight at 12 weeks
  HbA1c what value was stated as a percentage (%), were provided from participant's clinician before and 12 weeks after diet.
Amount of Fat mass | Change from Baseline Weight at 12 weeks
  Fat mass in kilograms was measured with TANİTA SC-330 instrument.
Rate of Body fat percentage | Change from Baseline Weight at 12 weeks
  Body fat percentage was calculated combined with weight and fat mass. Body fat percentage = (Body mass [kg] / Weight [kg]) x 100.
Amount of Fat free mass | Change from Baseline Weight at 12 weeks
  Fat free mass in kilograms, was measured with TANİTA SC-330 instrument.
Amount of Total body water | Change from Baseline Weight at 12 weeks
  Total body water in kilograms, was measured with TANİTA SC-330 instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Welton S, Minty R, O'Driscoll T, Willms H, Poirier D, Madden S, Kelly L. Intermittent fasting and weight loss: Systematic review. Can Fam Physician. 2020 Feb;66(2):117-125. PMID 32060194
- [Result] Rynders CA, Thomas EA, Zaman A, Pan Z, Catenacci VA, Melanson EL. Effectiveness of Intermittent Fasting and Time-Restricted Feeding Compared to Continuous Energy Restriction for Weight Loss. Nutrients. 2019 Oct 14;11(10):2442. doi: 10.3390/nu11102442. PMID 31614992
- [Result] Patterson RE, Sears DD. Metabolic Effects of Intermittent Fasting. Annu Rev Nutr. 2017 Aug 21;37:371-393. doi: 10.1146/annurev-nutr-071816-064634. Epub 2017 Jul 17. PMID 28715993
- [Result] Antoni R, Johnston KL, Collins AL, Robertson MD. Effects of intermittent fasting on glucose and lipid metabolism. Proc Nutr Soc. 2017 Aug;76(3):361-368. doi: 10.1017/S0029665116002986. Epub 2017 Jan 16. PMID 28091348